CLINICAL TRIAL: NCT05381363
Title: Inhaled Interferon α2b Treatment in Mild-to-moderate COVID-19 Infected Children
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: RenJi Hospital (Other); Shanghai Children's Hospital (Other); Shanghai Children's Medical Center, affiliated to Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHFudanU_COVID19-1
Record Dates: First submitted 2022-05-18; First posted 2022-05-19 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; Children
Keywords: interferon α2b; Inhaled treatment
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Inhaled Interferon α2b (Experimental): Inhaled Interferon α2b (10U/ml)
  Interventions: Drug: Inhaled Interferon α2b
- Intervention: Standard of Care (Other): Standard of care treatment will be provided according to management guideline.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Inhaled Interferon α2b — Drug: Inhaled Interferon α2b; 1-2 years old: 1 dose, three times per day; 3-7 years old: 1 dose, four times per day; 7-18 years old: 2 doses, four times per day
  Other Names: IFN α2b
  Arms: Intervention: Inhaled Interferon α2b
Other: Standard of Care — Standard of care treatment will be provided based on the New Coronavirus Pneumonia Prevention and Control guideline (9th edition), published by National Health Commission of China
  Other Names: SC
  Arms: Intervention: Standard of Care

SUMMARY:
In the COVID-19 pandemic era, a convenient and effective treatment for pediatric patients is unavailable. A multi-center Chinese clinical trials with the aim to using Interferon-α2b spray inhalation to develop new treatment strategies for the treatment of pediatric patients with mild or moderate type of COVID-19. The purpose of this study is to determine the safety and efficacy for Interferon α2b spray inhalation as first line treatment.

DETAILED DESCRIPTION:
This project aims to improve the treatment of pediatric patients infected with COVID-19. Interferon has antiviral property and is approved to be used in treatment in hepatitis B and hepatitis C virus infections. Interferon α2b, β1a and lambda are under evaluation in clinical trials for the treatment of COVID-19 in adult. As upper respiratory tract infection is the dominant characteristic of most infected children, topical treatment may be a better way to increase the safety and efficacy than oral or intravenous medication. This study aims to obtain essential data regarding the efficacy and safety of inhaled Interferon α2b in children with mild to moderate COVID-19 infection. Subjects will be enrolled with COVID-19 infection diagnoses by ORF1ab gene and N gene PCR test. Standard evaluation process will be applied to identify mild and moderate patients. Patients will be randomized into interferon group and non-interferon group. Patients in interferon group will receive inhalation treatment within the first five days since the symptom onset. Patients will receive daily PCR test. Cycle threshold (Ct) values over 35 is considered as de-isolation criterion. Days requiring isolation (from symptom onset to de-isolation time point) is the major index to evaluate efficacy. Clinical manifestations and test results from clinical recording system will be collected to evaluate the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as mild to moderate COVID-19 infection with positive PCR test and symptoms (Ct < 35)
* Parents and patients comprehend and welling to participate in this study.
* Agree to the collection of nasal swabs per day as protocol.

Exclusion Criteria:

* Patients evaluated as severe or critically severe type of COVID-19 infection (Individuals who have SpO2 <94% on room air, oxygen treatment is necessary, respiratory failure, septic shock, and/or multiple organ dysfunction).
* Patients with comorbidities
* Decline to participate by parents or children
* Allergy to any study medication or usage of any kind of interferon treatment within 14 days before test
* Children cannot tolerate the inhalation treatment
* Any situation where the program cannot be carried out safely.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Days requiring isolation (DRI) | from symptom onset to point of de-isolation (about 2-3 weeks)
  Efficacy of inhaled Interferon α2b by assessment of the Days requiring isolation (DRI). Patients will receive daily PCR. Nasal swab specimens were collected by standard procedures performed by trained nurses.

SECONDARY OUTCOMES:
Duration of fever | from fever onset to free from fever (about 2-3 weeks)
  Efficacy of inhaled Interferon α2b by assessment of the duration of fever.
Proportions of COVID-19 symptoms | from symptom onset to point of de-isolation (about 2-3 weeks)
  Efficacy of inhaled Interferon α2b by assessment of the duration of COVID-10 symptoms including fever, cough, sore throat, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell.
Blood test | Every 3 days (from the date of hospitalization to point of de-isolation)
  This test including the count of leukocytes, neutrophils, lymphocytes, platelets, and hemoglobin in plasma. Inflammatory Biomarker.
C-reactive protein (CRP) | Every 3 days (from the date of hospitalization to point of de-isolation)
  Inflammatory Biomarker
Interleukin 6 (IL-6) | Every 3 days (from the date of hospitalization to point of de-isolation)
  Inflammatory Biomarker
Chest imaging findings | once on admission
  Imaging evaluation methods
Number of Adverse Events (Abnormal Appearance) | From Day 1 to time point of de-isolation post-dose in each period (about 2-3 weeks)
  This is a composition of obviously severe flu-like symptoms, including nausea, fatigue, weight loss.
Number of Adverse Events (Abnormal Hematology) | From Day 1 to time point of de-isolation post-dose in each period (about 2-3 weeks)
  Safety of inhaled Interferon α2b by assessment of safety laboratory tests.
Number of Adverse Events (Abnormal Clinical Chemistry) | From Day 1 to time point of de-isolation post-dose in each period (about 2-3 weeks)
  Safety of inhaled Interferon α2b by assessment of safety laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramasamy S, Subbian S. Critical Determinants of Cytokine Storm and Type I Interferon Response in COVID-19 Pathogenesis. Clin Microbiol Rev. 2021 May 12;34(3):e00299-20. doi: 10.1128/CMR.00299-20. Print 2021 Jun 16. PMID 33980688
- [Background] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708
- [Background] Nile SH, Nile A, Qiu J, Li L, Jia X, Kai G. COVID-19: Pathogenesis, cytokine storm and therapeutic potential of interferons. Cytokine Growth Factor Rev. 2020 Jun;53:66-70. doi: 10.1016/j.cytogfr.2020.05.002. Epub 2020 May 7. PMID 32418715
- [Background] Zhou Q, Chen V, Shannon CP, Wei XS, Xiang X, Wang X, Wang ZH, Tebbutt SJ, Kollmann TR, Fish EN. Interferon-alpha2b Treatment for COVID-19. Front Immunol. 2020 May 15;11:1061. doi: 10.3389/fimmu.2020.01061. eCollection 2020. PMID 32574262
- [Background] Li C, Luo F, Liu C, Xiong N, Xu Z, Zhang W, Yang M, Wang Y, Liu D, Yu C, Zeng J, Zhang L, Li D, Liu Y, Feng M, Liu R, Mei J, Deng S, Zeng Z, He Y, Liu H, Shi Z, Duan M, Kang D, Liao J, Li W, Liu L. Effect of a genetically engineered interferon-alpha versus traditional interferon-alpha in the treatment of moderate-to-severe COVID-19: a randomised clinical trial. Ann Med. 2021 Dec;53(1):391-401. doi: 10.1080/07853890.2021.1890329. PMID 33620016
- [Background] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Background] Monk PD, Marsden RJ, Tear VJ, Brookes J, Batten TN, Mankowski M, Gabbay FJ, Davies DE, Holgate ST, Ho LP, Clark T, Djukanovic R, Wilkinson TMA; Inhaled Interferon Beta COVID-19 Study Group. Safety and efficacy of inhaled nebulised interferon beta-1a (SNG001) for treatment of SARS-CoV-2 infection: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Respir Med. 2021 Feb;9(2):196-206. doi: 10.1016/S2213-2600(20)30511-7. Epub 2020 Nov 12. PMID 33189161
- [Background] Mantlo E, Bukreyeva N, Maruyama J, Paessler S, Huang C. Antiviral activities of type I interferons to SARS-CoV-2 infection. Antiviral Res. 2020 Jul;179:104811. doi: 10.1016/j.antiviral.2020.104811. Epub 2020 Apr 29. PMID 32360182
- [Background] Zhou Q, MacArthur MR, He X, Wei X, Zarin P, Hanna BS, Wang ZH, Xiang X, Fish EN. Interferon-alpha2b Treatment for COVID-19 Is Associated with Improvements in Lung Abnormalities. Viruses. 2020 Dec 30;13(1):44. doi: 10.3390/v13010044. PMID 33396578
- [Background] Teraoka S, Sanaka T, Takahashi K, Toma H, Yamaguchi Y, Yagisawa T, Tanabe K, Sato H, Matsumura O, Nakajima I, et al. Stimulation of intrinsic prostacyclin synthesis and inhibition of thromboxane production to minimize cyclosporine nephrotoxicity. Transplant Proc. 1988 Jun;20(3 Suppl 3):638-45. No abstract available. PMID 3291300
- [Background] Hoagland DA, Moller R, Uhl SA, Oishi K, Frere J, Golynker I, Horiuchi S, Panis M, Blanco-Melo D, Sachs D, Arkun K, Lim JK, tenOever BR. Leveraging the antiviral type I interferon system as a first line of defense against SARS-CoV-2 pathogenicity. Immunity. 2021 Mar 9;54(3):557-570.e5. doi: 10.1016/j.immuni.2021.01.017. Epub 2021 Jan 29. PMID 33577760
- [Background] Kalil AC, Mehta AK, Patterson TF, Erdmann N, Gomez CA, Jain MK, Wolfe CR, Ruiz-Palacios GM, Kline S, Regalado Pineda J, Luetkemeyer AF, Harkins MS, Jackson PEH, Iovine NM, Tapson VF, Oh MD, Whitaker JA, Mularski RA, Paules CI, Ince D, Takasaki J, Sweeney DA, Sandkovsky U, Wyles DL, Hohmann E, Grimes KA, Grossberg R, Laguio-Vila M, Lambert AA, Lopez de Castilla D, Kim E, Larson L, Wan CR, Traenkner JJ, Ponce PO, Patterson JE, Goepfert PA, Sofarelli TA, Mocherla S, Ko ER, Ponce de Leon A, Doernberg SB, Atmar RL, Maves RC, Dangond F, Ferreira J, Green M, Makowski M, Bonnett T, Beresnev T, Ghazaryan V, Dempsey W, Nayak SU, Dodd L, Tomashek KM, Beigel JH; ACTT-3 study group members. Efficacy of interferon beta-1a plus remdesivir compared with remdesivir alone in hospitalised adults with COVID-19: a double-bind, randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Dec;9(12):1365-1376. doi: 10.1016/S2213-2600(21)00384-2. Epub 2021 Oct 18. PMID 34672949